CLINICAL TRIAL: NCT06774950
Title: Améliorer La Prise En Soins Et La Qualité De Vie Des Patients Diabétiques De Type 2 (Alliance DT2)
Brief Title: Value-based Care in Type 2 Diabetes (Enhancing T2D Care)
Acronym: Alliance DT2
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Réseau de soins Delta (Other)
Collaborators: University of St.Gallen (Other)
Responsible Party: Principal Investigator, Minette-Joëlle Zeukeng, Principal Investigator, Réseau de soins Delta
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2024-01350; SNCTP000006190 (Other: Swiss National Clinical Trials Portal)
Record Dates: First submitted 2024-12-10; First posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: The clinical trial has a complex trial design. The clinical trial is not a Decentralized Clinical Trials-DCT, nor has decentralized elements
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual care (No Intervention): Usual care
- Intervention arm (Experimental)
  Interventions: Behavioral: Physician-patient quality circle

INTERVENTIONS:
Behavioral: Physician-patient quality circle — Intervention: (To be compared with standard care)
  1. Interprofessionnal meeting per neighbourhood: (beforehand) Therapeutic patient education (TPE) training for healthcare professionals
  2. Physician-patient quality circle t0 Group sessions (n= 3 to 6 patients) with doctor and therapeutic patient education specialist Clinical measurements - CM (incl. HbA1c, body composition, blood pressure). PROM evaluation questionnaires (EQ5D&DIABQ)
  3. Development of individualised T2D programme: with case manager
  4. Quarterly follow-up: t3, t6, t9 months PROM follow-up (DIABQ&PHQ9) +CM.
  5. Evaluation of experience: t12 & t18 months PREM&PROM evaluation questionnaire +CM
  Arms: Intervention arm

SUMMARY:
The aim of this study is to obtain a better glycemic index score (decrease) by improving the care and quality of life of type 2 diabetic patients for a possible remission of diabetes.

This will be achieved through an intervention that includes a strategy for training primary care physicians and other healthcare professionals in patient therapeutic education (TPE), as well as group and/or individual TPE-related activities/tools made available to patients, funded and encouraged for individualized planning. Intervention follow-up will be carried out by means of quality-of-life questionnaires for patients who have undergone the new method, compared with patients who have received the usual care.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed type 2 diabetes (less than 10 years)
* Age (between 40 and 65)

Exclusion Criteria:

* Significant comorbidities linked to worsening diabetes (such as renal failure, previous myocardial infarction, retinopathy, signs or symptoms of severe diabetic neuropathy or diabetic foot ulcers), severe osteoarthritis or as judged by the attending physician.
* Pregnant or breast-feeding women
* Persons who are unable to give signed informed consent

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Glycated haemoglobin HbA1c (∆HbA1c) | During 18 month
  Mean change in glycated haemoglobin HbA1c (∆HbA1c)

SECONDARY OUTCOMES:
Health-related quality of life (∆ EQ-5D-5L) | During 18 months
  Mean change in health-related quality of life (∆ EQ-5D-5L). The EuroQol 5-Dimension 5-Level Health Questionnaire (EQ-5D-5L) scale measures health-related quality of life, including five dimensions, each rated on five levels. Utility scores range from -0.59 (negative scores are considered as worse than death) to 1.000 (perfect health), with higher scores indicating better health.
Diabetes self-care behaviours measured by the Diabetes Intention, Attitude, and Behavior Questionnaire (∆ DIAB-Q) | During 18 months
  Mean change in intention to adopt diabetes self-care behaviours (∆ DIAB-Q). Scores range from 0 (worst quality of life) to 100 (best quality of life), with higher scores indicating better outcomes and less impact of diabetes on daily life.
Fat/lean body mass (∆ body composition) | During 18 months
  Mean change in body fat/lean body mass (∆ body composition)
Cost-effectiveness analysis | At 12 and 18 months
  Cost-effectiveness analysis (∆HbA1c; costs assessed from the payer's point of view)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Geissler, PhD, Study Chair — University of St.Gallen

IPD SHARING:
Plan to Share IPD: Undecided
Depends on authorities

REFERENCES:
- [Derived] Ehlig D, Sapin M, Zeukeng MJ, Vogel J, Barthassat V, Favre B, DaCosta H, Tugay K, Coendoz-Carron S, Bumann D, Coclet J, Schaller P, Geissler A. Enhancing type 2 diabetes care by an individualized and group-based therapeutic patient education program: study protocol for a cluster randomized trial. Trials. 2025 Dec 23;26(1):577. doi: 10.1186/s13063-025-09302-x. PMID 41437100